CLINICAL TRIAL: NCT00438919
Title: The e-SELECT Registry a MULTICENTER POST-MARKET SURVEILLANCE
Brief Title: A Multi-center Post-Market Surveillance Registry
Acronym: E-SELECT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cordis US Corp. (Industry)
Responsible Party: Dr. Hans-Peter Stoll - Medical Affairs Director, Cordis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EC06-01
Record Dates: First submitted 2007-02-16; First posted 2007-02-22 (Estimated); Last update posted 2009-12-03 (Estimated); Status verified 2009-12

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Drug-Eluting Stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): CYPHER SELECT™ Sirolimus-eluting Coronary Stent
  Interventions: Device: drug-eluting stent

INTERVENTIONS:
Device: drug-eluting stent — CYPHER SELECT™ Sirolimus-eluting Coronary Stent

SUMMARY:
This multicenter, prospective, observational registry will evaluate the safety and performance of the CYPHER SELECT™ Sirolimus-eluting Coronary Stent, and of all future generation of commercially approved Cordis Sirolimus-eluting Stents (SES), in routine clinical practice. Its objective is to measure the incidence and identify the predictors of acute, sub-acute and late stent thrombosis and Major Adverse Cardiac Events (MACE). Additional analyses will be performed in patient sub-populations, such as diabetes, in-stent restenosis (ISR), acute myocardial infarction (AMI) and multivessel coronary disease.

DETAILED DESCRIPTION:
The data will be collected in consecutive subjects treated with commercially available product and following standard clinical practice. This registry will be limited to subjects who have received only the CYPHER SELECT™ Sirolimus-eluting Coronary Stent during the index procedure. While no inclusion or exclusion criteria have been specified, uniform, complete and accurate data will be collected peri-procedurally, during the index hospitalization, and during follow-up. All subjects should be treated according to the Instruction For Use (IFU) including conduct of the stenting procedure, application of antiplatelet medication and any other medical therapy should be provided according to local usual practice. Data collection (Electronic Data Capture), data management, statistical analyses, monitoring and core laboratory evaluations will be assigned to independent organizations.

ELIGIBILITY:
Inclusion Criteria:

* This registry will be limited to subjects who have received only the CYPHER SELECT™ Sirolimus-eluting Coronary Stent during the index procedure;
* Males and females;

Exclusion Criteria:

* None.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15000 (Estimated)
Dates: Start 2006-05; Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
acute, sub-acute and late stent thrombosis; Major Adverse Cardiac Events (MACE) | 1, 6, 12, 24 and 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Philip Urban, MD, Principal Investigator — Clinique La Tour
Locations (1):
- Clinique La Tour, Meyrin, Switzerland

REFERENCES:
- [Derived] Urban P, Abizaid A, Banning A, Bartorelli AL, Baux AC, Dzavik V, Ellis S, Gao R, Holmes D, Jeong MH, Legrand V, Neumann FJ, Nyakern M, Spaulding C, Worthley S; e-SELECT Investigators. Stent thrombosis and bleeding complications after implantation of sirolimus-eluting coronary stents in an unselected worldwide population: a report from the e-SELECT (Multi-Center Post-Market Surveillance) registry. J Am Coll Cardiol. 2011 Mar 29;57(13):1445-54. doi: 10.1016/j.jacc.2010.11.028. PMID 21435513